CLINICAL TRIAL: NCT06146283
Title: The Relationship Between Trunk Control and Hand Functions in Individuals With Parkinson's
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Nursena Kılıç, director, Sanko University
Other Study IDs: fztnursenakiliç
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Jamar Hydraulic Hand Dynamometer — This device measures hand grip strength. The individual should be in an upright sitting position. There should be no arm support on the sitting surface. ...
  The knee angle should be 90 degrees. Elbow angle should be 90 degrees. The wrist should be held without deviation. The measurement should be performed 3 times with an interval of 10 seconds.

SUMMARY:
The trunk, which plays an integral role in postural stabilization, controls extremity movements by providing dynamic stabilization during performance. Trunk stability is thought to be a prerequisite for upper extremity functions and it is assumed that trunk control has an effect on hand functions. There is thought to be a strong relationship between postural control and fine motor functions. There are very few studies in the literature examining the effect of trunk control on hand functions in Parkinson's patients. Based on this, the aim of this study is; To investigate the relationship between trunk control and hand functions.

* Hypotheses of the study;
* Ho: There is no relationship between Trunk Control and hand functions in individuals with Parkinson's disease.
* H1: There is a relationship between Trunk Control and hand functions in individuals with Parkinson's disease

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a progressive and neurodegenerative central nervous system disease characterized by loss of dopaminergic neurons in the substantia nigra. Rest tremor, bradykinesia, rigidity and postural instability are the four basic findings of Parkinson's disease. The progression of the disease varies from person to person, generally starting with unilateral findings, and after the third year, bilateral findings appear and progress from distal to proximal. Balance and postural control disorders also occur within two or three years. The first symptom seen in 80% of patients is rest tremor, which begins in the distal upper extremities. The trunk, which plays an integral role in postural stabilization, controls extremity movements by providing dynamic stabilization during performance. Trunk stability is thought to be a prerequisite for upper extremity functions and it is assumed that trunk control has an effect on hand functions. There is thought to be a strong relationship between postural control and fine motor functions. There are very few studies in the literature examining the effect of trunk control on hand functions in Parkinson's patients. Based on this, the aim of this study is; To investigate the relationship between trunk control and hand functions. Sociodemographic information will be recorded taking into account the answers to the questions in the personal information form prepared by the researcher. Parkinson's patients who meet the inclusion criteria; Rough Grip (Jamar Dynamometer), Nine Hole Peg Test (DDPT), Hoehn and Yahr Scale (HYÖ), Mini Mental Test, Quick-DASH, Duruöz Hand Index and Trunk Impairment Scale (GBÖ) will be performed by Physiotherapist Nursena KILIÇ.

As descriptive statistics; Mean and standard deviation or median and minimum-maximum values will be given for continuous variables specified by measurement, and frequency and percentage values will be given for qualitative variables. The suitability of continuous variables to normal distribution will be evaluated with the Kolmogorov-Smirnov test. In independent group comparisons; For continuous variables specified by measurement, if parametric test conditions are met, the significance test of the difference between two means or one-way ANOVA will be used. In cases where parametric test conditions are not met, Mann-Whitney U test or Kruskal-Wallis test will be used. In dependent measurement comparisons, the significance test of the difference between two pairs will be used for normally distributed data, and the Wilcoxon paired two sample test will be used for non-normally distributed data. The relationship between two continuous variables will be evaluated with Pearson or Spearman Rank correlation coefficients. p<0.05 was considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 40 and 70,
* Being diagnosed with Parkinson's disease by a neurologist,
* Having a Mini Mental Test score of 24 and above,
* Modified Hoehn Yahr Scale score is 2 or less than 2,
* Having no additional neurological or orthopedic disease

Exclusion Criteria:

* Individuals with advanced cognitive problems and aphasia,
* Individuals with additional neurological disorders,
* Individuals who refuse to participate in the study,
* Individuals with vision and hearing problems will not be included.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included individuals diagnosed with Parkinson's between the ages of 40-70.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Nine Hole Peg Test (9DPT) | 1 weeks
  Nine Hole Peg Test (9DPT): It is a valid and reliable skill test frequently used to evaluate upper extremity function.
Hand Grip Strength Measurement | 1 weeks
  Hand Grip Strength Measurement: It is recommended by the American Association of Hand Therapists (AETD) for measuring hand grip strength and has been found to have high validity and reliability in many studies and is therefore considered the gold standard.
Hoehn and Yahr Scale (HYS) | 1 weeks
  Hoehn and Yahr Scale (HYS):t is a staging system developed by Hoehn and Yahr that provides information in a short time in determining the degree and symptoms of the disease in individuals with Parkinson's disease. The scale value is between 1-5
Mini Mental Test (MMT) | 1 weeks
  Mini Mental Test (MMT):The test was produced as a cognitive assessment tool that takes a short time to apply in the examination of the elderly, especially the elderly with delirium and/or dementia, since the tests used to quantitatively evaluate cognitive performance within standard neuropsychiatric examination methods contain too many questions and take more than 30 minutes to apply.
Quick-DASH | 1 weeks
  Quick-DASH:It is an evaluation questionnaire that measures activity and participation limitations in all upper extremity disorders. In the survey, patients' difficulties during daily living activities are questioned with 11 questions. Each question has 5 answer options according to difficulty level. If the patient can do the activity without difficulty, he/she marks 1, if he/she has mild difficulty, 2, if he/she has moderate difficulty, 3, if he/she has extreme difficulty, 4, and if he/she cannot do it at all, he/she marks option 5.
Duruöz Hand Index | 1 weeks
  Duruöz Hand Index:It consists of 18 questions filled out by patients to evaluate hand disability. This scale includes questions divided into 5 categories: kitchen chores, dressing, personal hygiene, workplace and other activities. Answers are scored as: I don't have difficulty (=0), I have little difficulty (=1), I have some difficulty (=2), I have great difficulty (=3), it is almost impossible to do it (=4), I definitely cannot do it (=5). The total score consists of the sum of all scores. (0-90). High scores indicate impaired hand functions
Trunk Impairment Scale | 1 weeks
  Trunk Impairment Scale:This scale consists of three subscales; static-dynamic sitting balance and trunk coordination. GDS value varies between 0-23 and a high score indicates good trunk control.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided